CLINICAL TRIAL: NCT02003547
Title: A Single Centre, Placebo-Controlled, Double-Masked, Sequential Designed Study to Evaluate 3 Ophthalmic Formulations of AMA0076 in Healthy Subjects
Brief Title: A Single Centre Study to Evaluate 3 Ophthalmic Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amakem, NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMA0076-M-101; 2013-002334-21 (EudraCT Number)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma; Ocular Hypertension; Eye Disease
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AMA0076 Formulation A (Experimental): Topical Ocular Drop BID X 1 wk
  Interventions: Drug: AMA0076
- AMA0076 Formulation B (Experimental): Topical Ocular Drop BID X 1wk
  Interventions: Drug: AMA0076
- AMA0076 Formulation C (Experimental): Topical Ocular Drop BID X 1 wk
  Interventions: Drug: AMA0076
- Placebo (Placebo Comparator): Topical Ocular Drop BID X 1 wk
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMA0076
  Arms: AMA0076 Formulation A; AMA0076 Formulation B; AMA0076 Formulation C
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Single Centre, Placebo-Controlled, Double-Masked, Sequential Designed Study to Evaluate 3 Ophthalmic Formulations of AMA0076 in Healthy Subjects

DETAILED DESCRIPTION:
Each subject will receive the following treatments:

* Period 1: Formulation A (n = 14) or placebo (n = 7) twice daily for 7 days
* Period 2: Formulation B (n = 14) or placebo (n = 7) twice daily for 7 days
* Period 3: Formulation C (n = 14) or placebo (n = 7) twice daily for 7 days

There will be a minimum washout of 7 days between each treatment period (last dose of previous period to first dose of subsequent period

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant, non-lactating females, aged 35 to 65 years.
* Body mass index of ≤35kg/m2.
* IOP between 15 and 24 mmHg (inclusive) in both eyes at Screening Visits 1 and 2.

Exclusion Criteria:

* Women of child-bearing potential who have a positive pregnancy test.
* Any subject deemed by the investigator to have uncontrolled systemic hypertension
* Use of systemic, inhaled or ocular corticosteroid treatment within 90 days of screening or likely to require their use during the study period.
* Any screening laboratory abnormality that, in either the investigator's or the medical monitor's judgment, is considered to be clinically significant or a safety risk.
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results of the subject's ability to participate in the study, or interfere with interpretation of the subject's study results.
* Participation in any other clinical study within 1 month of screening or during the study.
* Receipt of another investigational drug within 90 days of dosing in this study
* Diagnosis of any form of glaucoma.
* IOP >24 mmHg in either eye at any screening visit.
* Use of any ocular drops (including lubricating drops/artificial tears) during screening period or need for ocular drops during duration of study participation.
* In the opinion of the investigator, clinically significant eye trauma within 6 months of screening.
* Any intraocular ophthalmic procedure within 6 months of screening.
* Any ocular inflammation within 90 days of screening or a history of recurrent uveitis in either eye.
* Subjects with any known ocular disease and who are under care of a hospital ophthalmologist.
* Any condition preventing valid applanation tonometry measurement.
* Unable to discontinue contact lens wear during the study
* Visual acuity (VA) worse than 20/80 in either eye
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
* History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption.
* Positive drugs of abuse test result.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 7 days
  The primary endpoint is the comparison of Intraocular Pressure assessments taken at pre-treatment on Day -1 and on Day 7 for each diurnal time point (0, 2, 4 and 8 h post-anticipated dose [Day -1] or post-dose [Day 7]) for each treatment period between active treatment and placebo.

SECONDARY OUTCOMES:
Safety and Tolerability | 7 days
  The secondary endpoints are:
  * Comparison of hyperaemia assessments in each eye using a photographic rating scale on Day -1 (0 and 8 h post-anticipated dose) and Day 7 (0, 2, 4 and 8 h post dose)
  * Assessment of ocular surface photographic images of each eye on Day -1 and Day 7 (0 h).
  * Safety laboratory assessments, vital signs, 12-lead electrocardiogram (ECG), recording of Adverse Events and ophthalmic examination findings including visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, Principal Investigator — Quotient Clinical
Locations (1):
- Ruddington, Nottingham, United Kingdom